CLINICAL TRIAL: NCT07060014
Title: Liposomal Irinotecan (Nal-IRI) Plus 5-fluorouracil and Leucovorin (5-FU/LV) Plus Oxaliplatin (NALIRIFOX) as First-Line Chemotherapy for Patients With Advanced Small Intestine and Appendiceal Cancers
Brief Title: NALIRIFOX (Nal-IRI Plus 5-FU/LV Plus Oxaliplatin) as First-Line Treatment for Patients With Advanced Small Intestine and Appendiceal Cancers
Status: Not yet recruiting | Phase: Phase 1 | Type: Interventional
Sponsor: The Methodist Hospital Research Institute (Other)
Responsible Party: Principal Investigator, Maen Abdelrahim, MD, PhD, Pharm.B, Chief Gastrointestinal Medical Oncology, The Methodist Hospital Research Institute
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: PRO00038285
Record Dates: First submitted 2025-06-10; First posted 2025-07-11 (Actual); Last update posted 2025-07-11 (Actual); Status verified 2025-06

CONDITIONS: Advanced Small Intestine Cancer; Appendiceal Cancers
Keywords: Advanced Small Intestine cancer; Appendiceal Cancers
MeSH Terms: interventions — irinotecan sucrosofate; Fluorouracil; Oxaliplatin

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: No

ARMS (2):
- nal-IRI plus 5-FU/LV plus NALIRIFOX (Experimental): Patients in this arm will receive NALIRIFOX
  Interventions: Drug: Patients will be treated with NALIRIFOX (liposomal irinotecan 50 mg/m2 + 5-FU 2400 mg/m2 + LV 400 mg/m2 + oxaliplatin 60 mg/m2, IV) every 2 weeks for 12 months
- Historical Control Arm (No Intervention)

INTERVENTIONS:
Drug: Patients will be treated with NALIRIFOX (liposomal irinotecan 50 mg/m2 + 5-FU 2400 mg/m2 + LV 400 mg/m2 + oxaliplatin 60 mg/m2, IV) every 2 weeks for 12 months — The study drugs will be administered per the regimen defined in the NAPOLI-3 clinical trial. Patients will be treated with NALIRIFOX (liposomal irinotecan 50 mg/m2 + 5-FU 2400 mg/m2 + LV 400 mg/m2 + oxaliplatin 60 mg/m2, IV) every 2 weeks for 12 months.
  Arms: nal-IRI plus 5-FU/LV plus NALIRIFOX

SUMMARY:
This study will evaluate the safety and efficacy of NALIRIFOX per NAPOLI-3 regimen as first-line chemotherapy for patients with advanced small intestine and appendiceal cancers. Female or male patients aged 18 years, or older, with histopathologically or cytologically confirmed advanced mucinous or non-mucinous appendix cancer or advanced small intestine cancer will be eligible for participation in the study.

DETAILED DESCRIPTION:
This study will evaluate the safety and efficacy of NALIRIFOX per NAPOLI-3 regimen as first-line chemotherapy for patients with advanced small intestine and appendiceal cancers. Female or male patients aged 18 years, or older, with histopathologically or cytologically confirmed advanced mucinous or non-mucinous appendix cancer or advanced small intestine cancer will be eligible for participation in the study. Approximately, 22 patients will be enrolled in the study. The study drugs will be administered per the regimen defined in the NAPOLI-3 clinical trial, NCT04083235. Patients will be treated with NALIRIFOX (liposomal irinotecan 50 mg/m2 + 5-FU 2400 mg/m2 + LV 400 mg/m2 + oxaliplatin 60 mg/m2) every 2 weeks for 12 months.

ELIGIBILITY:
Inclusion Criteria:

1. Male or female ≥18 years of age.
2. Histopathologically or cytologically confirmed advanced mucinous or non-mucinous appendix cancer or advanced small intestine cancer.
3. Measurable disease per the Response Evaluation Criteria in Solid Tumors (RECIST) v1.1.
4. Eastern Cooperative Oncology Group performance status of 0 or 1.
5. Life expectancy ≥6 months.
6. Patients of childbearing potential must agree to use an adequate method of contraception during the study and for 30 days after the last dose of study treatment.

Exclusion Criteria:

* 1. Hematology laboratory values of:

  1. Absolute neutrophil count ≤1500 cells/mm3
  2. Platelets ≤100,000 cells/mm3
  3. Hemoglobin ≤9 g/dL
  4. White blood count ≤3000 cells/mm3. 2. Hepatic laboratory values of aspartate transaminase or alanine aminotransferase:

  <!-- -->

  1. >5 × upper limits of normal (ULN) if the documented history of hepatic metastases; or
  2. >2.5 × ULN if no liver metastases are present. 3. Total bilirubin >1.5 × ULN or >1.5 mg/dL. 4. Prothrombin time (PT) or international normalized ratio (INR) >1.5 × ULN. Note: Patients receiving therapeutic doses of anticoagulant therapy may be considered eligible if PT and INR are within the acceptable institutional therapeutic limits.

     5. Serum creatinine or serum urea >1.5 × ULN. 6. Estimated glomerular filtration rate <50 mL/min. 7. Positive pregnancy test, pregnancy, or breastfeeding (female patients only). 8. Any other clinically significant laboratory abnormality that would compromise patient safety or the outcome of the study.

     9. Any clinically significant and/or uncontrolled cardiac-related abnormality that would compromise patient safety or the outcome of the study including, but not limited to:

  <!-- -->

  1. Arrhythmia
  2. Bradycardia
  3. Tachycardia
  4. Symptomatic valvular disease
  5. Symptomatic congestive heart failure is classified by the New York Heart Association as Class III or IV
  6. Unstable angina pectoris. 10. Myocardial infarction within the past 6 months. 11. Active bleeding diathesis. 12. Current complaints of persistent constipation or history of chronic constipation, bowel obstruction, or fecaloma within the past 6 months.

     13. Receiving chronic treatment with corticosteroids ≥5 mg of prednisone per day (or equivalent) or another immunosuppressive agent (s) 14. Known history and/or uncontrolled hepatitis B surface antigen, hepatitis C antibody, or human immunodeficiency virus (HIV)-1 or HIV-2.

     15. History of galactose intolerance, deficiency of Lapp lactase, or glucose-galactose malabsorption.

     16. History of malignancy or active treatment for malignancy (i.e., radiation or chemotherapy, including monoclonal antibodies) within 5 years. Note: Patients with squamous or basal cell carcinomas of the skin, carcinomas in situ of the cervix or uterus, ductal breast cancer in situ, resected low-grade prostate cancer, or other malignancies that in the opinion of the investigator are considered cured may participate.

     17. Receipt of live, attenuated vaccine (e.g., intranasal influenza, measles, mumps, rubella, varicella) or close contact with someone who has received a live, attenuated vaccine within the past 1 month. Note: Influenza vaccine will be allowed if administered >21 days.

     18. Receipt of any investigational agent or study treatment within the past 30 days.

     19. Receipt of any protein or antibody-based therapeutic agents (e.g., growth hormones or monoclonal antibodies) within the past 3 months.

     20. Allergies reaction to irinotecan or liposomal irinotecan.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 22 (Estimated)
Dates: Start 2025-07-18 (Estimated); Primary Completion 2026-09-30 (Estimated); Study Completion 2026-12-31 (Estimated)

PRIMARY OUTCOMES:
Number of participants with treatment-related adverse events as assessed by CTCAE v5.0 in patients receiving Nalirifox per Napoli-3 regimen as first-line chemotherapy for advanced non-resectable small intestine and appendiceal cancers | Over 12 months
  This measure evaluates the safety and tolerability of Nalirifox per Napoli-3 regimen by reporting the number of participants experiencing treatment-related adverse events, graded according to the Common Terminology Criteria for Adverse Events (CTCAE) version 5.0. Data will be collected through clinical assessments, including physical examinations, laboratory tests, and patient-reported adverse events, and summarized as the total count and severity of events per participant.

SECONDARY OUTCOMES:
Duration of response to Nalirifox per Napoli-3 regimen as first-line chemotherapy in patients with advanced non-resectable small intestine and appendiceal cancers, assessed by RECIST v1.1 | Over 12 months
  This measure evaluates the duration of response to Nalirifox per Napoli-3 regimen, defined as the time from the first documented objective response (complete response or partial response) per Response Evaluation Criteria In Solid Tumors (RECIST) v1.1 until disease progression or death, whichever occurs first. Data will be collected through radiographic assessments (e.g., CT or MRI scans) at regular intervals and summarized as the median duration of response in months.

CONTACTS AND LOCATIONS:
Overall Officials: Abdullah Esmail, MD, Study Director — Houston Methodist Nael Cancer Center
Locations (1):
- Houston Methodist Hospital, Houston, Texas, United States

IPD SHARING:
Plan to Share IPD: No